CLINICAL TRIAL: NCT04103320
Title: Evaluation of Pain in the Course of in Vitro Fertilization: the Endalgofiv Study
Brief Title: Evaluation of Pain in the Course of in Vitro Fertilization
Acronym: ENDALGOFIV
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_45; 2019-A00555-52 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-08-28; First posted 2019-09-25 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Infertility
Keywords: Infertility; In Vitro Fertilization; Endometriosis; pain evaluation
MeSH Terms: conditions — Infertility; Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Using different survey to evaluate pain — Survey will be at different time of the IVF protocol (at the first medical appointment in the medically assisted department, after stimulation, after oocytes retrieval, after embryo transfer, one month after the IVF protocol)

SUMMARY:
25 to 50% of endometriotic patients are infertile and use medically assisted procreation. In general, the assessment of pain in medically assisted procreation is very little studied. Pain assessment studies in endometriotic patients remain limited to a quantitative assessment of pain symptomatology, without contextualization of painful manifestations. The primary objective of our study is the qualitative and contextualized assessment of pain during In Vitro Fertilization (IVF) protocol in endometriotic and non-endometriotic patients. The secondary objectives of our study are the quantitative study of pain, the measurement of the impact of personal efficiency on painful symptomatology, evaluation of depression, the results of IVF (implantation, pregnancy and live birth rates), and compare pain between endometriotic or non-endometriotic patients and between primary infertility and secondary infertility. According to the results obtained in this study, therapeutic strategies for the management of pain could be proposed, with the aim of improving the quality of life and the results of IVF in these patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients who start an IVF cycle in the medically assisted procreation department of the Jeanne de Flandres Hospital (CHRU Lille)

Exclusion Criteria:

* Refusal to participate in the study
* Minor patient
* Patient over 43 years old
* BMI patient > 35
* Pregnant woman
* Unable to provide clear information to the patient
* Patient under guardianship or lack of health cover
* Patient in IVF with donation of oocyte
* IVF patients for oocyte preservation
* Patient who had already participated in the study

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All patients who start an IVF cycle in the medically assisted procreation department of the Jeanne de Flandres Hospital (CHRU Lille)
Study Population: All patients who start an IVF cycle in the medically assisted procreation department of the Jeanne de Flandre Hospital (CHRU Lille)
Sampling Method: Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Comparison of the scores obtained by the pain survey (EN, QDSA, DN4), quality of life survey (EQ-5D), depression and anxiety (HAD), pain catastrophism score (PCS) and assessment of personal efficacy (heiQ). | one month after the IVF protocol
  composite criteria to assess of the typology of pain
EN = numerical scale of pain | one month after the IVF protocol
  from 0 to 10 (0 is "no pain" and 10 is "maximum pain imaginable")
Questionnaire douleur Saint Antoine (QDSA) | one month after the IVF protocol
  QDSA for emotional and sensory dimension of pain. It's a word list to describe a pain, patient must specify the type of pain that she usually feels for 8 days by putting a cross for the correct answer (0 to 4: absent, weak, moderate, strong, extremely strong)
DN4 | one month after the IVF protocol
  emotional and sensory dimension of pain, neuropathic pain survey in four questions - score on 7
EQ-5D quality of life | one month after the IVF protocol
  overall score on a numeric scale "check the box that best describes your health today", 5 themes (mobility, autonomy of the person, common activities, pain / discomfort, anxiety / depression)
HAD,anxiety and depression | one month after the IVF protocol
  2 scores on 21 - "circle the number that best fits your condition"
pain catastrophism scale (PCS) | one month after the IVF protocol
  score between 0 to 52
heiQ = personal efficiency, | one month after the IVF protocol
  40 questions with 8 dimensions

SECONDARY OUTCOMES:
Comparison of the scores obtained by the pain survey (EN, QDSA, DN4), quality of life survey (EQ-5D), depression and anxiety (HAD), pain catastrophism score (PCS) and assessment of personal efficacy (heiQ). | at Baseline (the first medical appointment) and 15 days after the embryo transfer
  composite criteria to assess of the typology of pain
implantation rates (%) | at Baseline (the first medical appointment), 15 days after embryo transfer, and at one month of the IVF cycle
  measure in endometriotic and non-endometriotic patients,in primary and secondary infertility patients
pregnancy rate (%) | at Baseline (the first medical appointment), 15 days after embryo transfer, and at one month of the IVF cycle
  measure in endometriotic and non-endometriotic patients,in primary and secondary infertility patients
live birth rate (0 or 1) | at Baseline (the first medical appointment), 15 days after embryo transfer, and at one month of the IVF cycle
  measure in endometriotic and non-endometriotic patients,in primary and secondary infertility patients
renouncing a new IVF attempt: yes or no | at Baseline (the first medical appointment), 15 days after embryo transfer, and at one month of the IVF cycle
  measure the impact of pain on the pregnancy project in endometriotic and non-endometriotic patients,in primary and secondary infertility patients
willingness to take a specific treatment with an analgesic goal: yes or no answer | at Baseline (the first medical appointment), 15 days after embryo transfer, and at one month of the IVF cycle
  measure the impact of pain on the pregnancy project in endometriotic and non-endometriotic patients,in primary and secondary infertility patients

CONTACTS AND LOCATIONS:
Overall Officials: Chrystelle Rubod, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France